CLINICAL TRIAL: NCT02220582
Title: A Pan-Canadian, Multi-ethnic Cohort Study in Healthy Participants Aimed to Better Understand the Impact of Individual, Socioeconomic and Other Environmental Factors Leading to Cardiac and Vascular Disease
Brief Title: Canadian Alliance for Healthy Hearts and Minds
Status: Completed | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CAHHM
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiac Magnetic Resonance (CMR); Cardiovascular Diseases; socio-environmental factors; Contextual factors
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study will precisely phenotype individuals with respect to cardiac, vascular and cognitive dysfunction and to identify novel targets for indicators of early disease.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: MRI — Magnetic Resonance Imaging

SUMMARY:
The Cardiac, Vascular and Cognitive Dysfunction (CVCD) Alliance will be a prospective, multi-ethnic cohort study in healthy Canadian individuals between 35 and 69, looking at contextual risk factors and novel predictors of hard events over a period of four years.

The unique features of this initiative are:

* MRI as the sole imaging technique (including the use of a mobile MRI machine)
* Contextual factor analysis (including community environmental profile assessments)
* Record linkage follow-up of individuals to health services (administrative) databases for major morbidity and mortality events and health services utilization

DETAILED DESCRIPTION:
Cardiac, vascular, and cognitive dysfunction have a strong impact on the quality of life, longevity and health care costs, in Canada and globally. Cardiovascular risk factors account for up to half of the attributable risk for dementia, mediated in large part by difficult to detect microvascular disease of the brain. In this study the investigators will try to understand the role of the societal structure, nutrition, access to health services, and other socio-environmental and contextual factors on cardiovascular risk factors, subclinical disease and clinical cardiovascular events at the individual and population levels. We will try to identify markers for early subclinical dysfunction in the brain, vessels, heart and abdomen using magnetic resonance imaging and investigate the associations with contextual and individual determinants of these markers, as well as to assess the predictive value of novel markers of subclinical dysfunction on the development of clinical cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Form (ICF) was discussed, understood and signed by the participant
* Participant is between ages 35 and 69 (inclusively) at time of screening
* The participant is willing to undergo an MRI scan and all other required study procedures

Exclusion Criteria:

* Participant has a known acute disease or condition that is considered serious in the investigator's opinion
* Participant is claustrophobic and/or is known to suffer from moderate to severe anxiety during MRI scans or similar procedures
* Participant is obese and/or exceeds equipment weight limit and/or circumference of the MRI portal at this of screening
* Participant has any kind of metallic device that would contra-indicate Magnetic Resonance Imaging (MRI) (e.g. pacemakers, defibrillator, vascular clips, drug pumps, implant(s), or any other foreign bodies)
* Participant has an extensive tattoo covering a large part of their chest or head
* Female participants that are currently pregnant (confirmed or uncertain).
* Participants receiving Gadovist® only - Female participants that are currently breastfeeding.
* Participants receiving Gadovist® only - Participant has a known hypersensitivity to gadolinium-based contrast agents
* Participants receiving Gadovist® only - Participant has a known allergy or severe reaction to any contrast agent typically used in MRI procedures
* Participants receiving Gadovist® only - Participant has known renal or hepatic impairment of any intensity or any other kidney/liver disease or has recently undergone kidney/liver transplant
* Participants receiving Gadovist® only - Participant has a known glomerular filtration rate (eGFR or GFR) of 30 mL/min or less
* Participants receiving Gadovist® only - Participant has taken part in a clinical research study or clinical study within 30 days prior to enrollment in this study, and/or received contrast agent within 72 hours prior to the study MRI

Ages: 35 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants of Canadian Partnership for Tomorrow Project (CPTP) cohorts (BC Generations, Alberta Tomorrow Project, Ontario Health Study, CARTaGENE, Atlantic PATH) or non--CPTP cohorts (Montreal Heart Institute Biobank or the Prospective Urban-Rural Epidemiology, PURE study, or aboriginal cohort participants).
  Multi-ethnic participants including reserve-based Aboriginal peoples.
Sampling Method: Non-Probability Sample
Enrollment: 7900 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Myocardial Infarction (MI) | After completion of MRI and during follow-up period (2 to 3 years)
Stroke | After completion of MRI and during follow-up period (2 to 3 years)
Percutaneous Transluminal Coronary Angioplasty | After completion of MRI and during follow-up period (2 to 3 years)
Percutaneous Coronary Intervention | After completion of MRI and during follow-up period (2 to 3 years)
Coronary Artery Bypass Graft | After completion of MRI and during follow-up period (2 to 3 years)

SECONDARY OUTCOMES:
Congestive Heart Failure | After completion of MRI and during follow-up period (2 to 3 years)
  Congestive Heart Failure requiring hospitalization
New onset established risk factors | After completion of MRI and during follow-up period (2 to 3 years)
  * Incident diagnosis of diabetes by physician
  * Incident diagnosis of arterial hypertension by physician
  * Incident diagnosis of significant cognitive dysfunction (i.e. dementia) by physician.
Risk markers acquired through imaging and blood samples | After completion of MRI and during follow-up period (2 to 3 years)
  * Acquired parameters that are linked to the present health status
  * Candidate parameters for predicting cardiovascular events which affect cardiac and cognitive dysfunction. For further details, please see list of outcomes in the questionnaires and the MRI protocol described in section 4 above

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Friedrich, MD, Principal Investigator — Montreal Heart Institute; Sonia Anand, PhD, Principal Investigator — McMaster University; Jack Tu, MD, Principal Investigator — Institute for Clinical Evaluative Sciences
Locations (12):
- Canada (12):
  - Seaman Family MR Research Center, Calgary, Alberta
  - University of Calgary, Calgary, Alberta
  - St Paul's Hospital, Vancouver, British Columbia
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Robarts Research Institute, London, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Montreal Heart Insitute, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - IUCPQ, Ste Foy, Quebec

REFERENCES:
- [Derived] Luu JM, Gebhard C, Ramasundarahettige C, Desai D, Schulze K, Marcotte F, Awadalla P, Broet P, Dummer T, Hicks J, Larose E, Moody A, Smith EE, Tardif JC, Teixeira T, Teo KK, Vena J, Lee DS, Anand SS, Friedrich MG; CAHHM Study Investigators. Normal sex and age-specific parameters in a multi-ethnic population: a cardiovascular magnetic resonance study of the Canadian Alliance for Healthy Hearts and Minds cohort. J Cardiovasc Magn Reson. 2022 Jan 3;24(1):2. doi: 10.1186/s12968-021-00819-z. PMID 34980185
- [Derived] Luu JM, Sergeant AK, Anand SS, Desai D, Schulze K, Knoppers BM, Zawati MH, Smith EE, Moody AR, Black SE, Larose E, Marcotte F, Kleiderman E, Tardif JC, Lee DS, Friedrich MG; CAHHM Study Investigators. The impact of reporting magnetic resonance imaging incidental findings in the Canadian alliance for healthy hearts and minds cohort. BMC Med Ethics. 2021 Oct 28;22(1):145. doi: 10.1186/s12910-021-00706-3. PMID 34711210
- [Derived] Teixeira T, Hafyane T, Stikov N, Akdeniz C, Greiser A, Friedrich MG. Comparison of different cardiovascular magnetic resonance sequences for native myocardial T1 mapping at 3T. J Cardiovasc Magn Reson. 2016 Oct 4;18(1):65. doi: 10.1186/s12968-016-0286-6. PMID 27716344